CLINICAL TRIAL: NCT02377908
Title: European Postgraduate Training in Geriatric Medicine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Klinikum Nürnberg (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Principal Investigator, PD Dr. Katrin Singler, MME, Medical Doctor, Klinikum Nürnberg
Other Study IDs: KS-RRW EU survey
Record Dates: First submitted 2015-02-17; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Education; Geriatrics

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Online Survey — Online questionaire submitted to experts in geriatrics in different European countries. 12-item survey.

SUMMARY:
The objective of the study is to give a structured update on geriatric postgraduate education throughout Europe. The study will be performed as a cross-sectional structured quantitative online survey with qualitative comments. The survey content covers structural items, content and educational aspects of geriatric specialty training in European countries.

DETAILED DESCRIPTION:
The study is performed as a cross-sectional structured quantitative survey leaving space for qualitative comments. The survey content covers structural items, content and educational aspects of geriatric specialty training in European countries. To prove feasibility in the questionnaire setting and time management the survey will be piloted in five international experts in geriatric medicine. Questions in the survey are closed with the possibility to give a free comment.Validity of individual data collection will be controlled by repeated hidden content within different questions.

Experts in the field of geriatric medicine and members of one of the organizations European Union of Medical Specialists (UEMS), European Academy for the Medicine of Ageing (EAMA) or European Union Geriatric Medicine Society (EUGMS) and a strong personal focus of interest in postgraduate training are contacted by the survey coordinator and invited to participate in the survey personally and via E-mail. The survey will be performed online using the following software (http://www.surveyxact.com/) . To reassure data quality, the survey will be sent for double checks within nations.

ELIGIBILITY:
Inclusion Criteria:

Experts in geriatric medicine and member of one of the organizations European Union of Medical Specialists (UEMS), European Academy for the Medicine of Ageing (EAMA) or European Union Geriatric Medicine Society (EUGMS).

Exclusion Criteria:

none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Experts in geriatric medicine and member of one of the organizations European Union of Medical Specialists (UEMS), European Academy for the Medicine of Ageing (EAMA) or European Union Geriatric Medicine Society (EUGMS).
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
situation of geriatric postgraduate education | until June 2014
  Evaluate a structured update on geriatric postgraduate education throughout Europe in order to assess the need for further developments in geriatric postgraduate education.

CONTACTS AND LOCATIONS:
Locations (1):
- Insitute for Biomedicine of Aging, Nuremberg, Bavaria, Germany